CLINICAL TRIAL: NCT00468026
Title: Evaluation of the ProstaPlant Prostate Stent Insertion in Ex Vivo Human Prostate
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ProstaPlant Urology System Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Human Ex-Vivo - V001-3.2007
Record Dates: First submitted 2007-04-30; First posted 2007-05-01 (Estimated); Last update posted 2007-05-01 (Estimated); Status verified 2007-03

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH; Prostate; Stent; Benign prostatic hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

INTERVENTIONS:
Device: ProstaPlant Stent

SUMMARY:
The purpose of this ex-vivo study is to evaluate the insertion procedure for the ProstaPlant implant in human prostates and the support that it supplies to the prostate.

ELIGIBILITY:
Inclusion Criteria:

* Males,
* 18 years old and up,
* Suffer from BPH,
* Candidate for radical prostatectomies

Exclusion Criteria:

* According to the physician's decision

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
This is a feasibility study, in which initial evaluation of stent insertion procedure is obtained

CONTACTS AND LOCATIONS:
Overall Officials: Jack Baniel, Prof., Principal Investigator — "Rabin" Medical Center - "Belinson" Campus - Urology Department
Locations (1):
- "Asuta" Medical Center, Tel Aviv, Israel